CLINICAL TRIAL: NCT04684381
Title: A Phase 4, Open-Label, Single-Center Study to Assess Pharmacokinetic Characteristics and Safety of Endari in Patients With Sickle Cell Disease
Brief Title: Pharmacokinetics and Safety of Endari (L-glutamine) in Sickle Cell Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emmaus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EM-PK-01
Record Dates: First submitted 2020-12-18; First posted 2020-12-24 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Sickle Cell Disease; Pharmacokinetics
Keywords: Sickle cell disease; pharmacokinetics; L-glutamine
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- L-glutamine (Experimental): Pharmacokinetic characteristics of L-glutamine
  Interventions: Drug: L-glutamine

INTERVENTIONS:
Drug: L-glutamine — Pharmacokinetic study
  Other Names: Endari

SUMMARY:
L-glutamine has been approved in the US to reduce the acute complications of sickle cell disease (SCD) in adult and pediatric patients 5 years of age and older. The purpose of this single-center, open-label, phase 4 study is to evaluate the pharmacokinetic characteristics and safety of L-glutamine in patients with SCD.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is associated with a mutation in the β-hemoglobin gene that results in abnormal polymerization of hemoglobin. Polymerization of hemoglobin causes the red blood cell to sickle, leading to a cascade of events which cause acute complications for SCD patients.

L-glutamine has been approved in the US to reduce the acute complications of sickle cell disease (SCD) in adult and pediatric patients 5 years of age and older.

The purpose of this single-center, open-label, phase 4 study is to evaluate the pharmacokinetic characteristics and safety of L-glutamine in patients with SCD.

8 SCD patients and 4 healthy volunteers will receive weight-based dosing of L-glutamine for 3 weeks. Doses will be changed weekly: 0.1 g/kg administered twice daily during week 1, 0.3 g/kg administered twice daily during week 2, and 0.6 g/kg administered once daily during week 3.

The primary objective is to evaluate the pharmacokinetic characteristics of L-glutamine in SCD patients compared with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. 5 years of age and older at Screening.
2. Has documented diagnosis of SCD with known genotype (HbSS, HbSβ0 and HbSC).
3. Written informed consent provided by patient or the patient's legally authorized representative.
4. Non-pregnant females of childbearing age must agree to avoid pregnancy during the study and to practice a recognized form of birth control during the course of the study (e.g., barrier, birth control pills, or abstinence).

Inclusion Criteria for Healthy Volunteers:

1. No known hematologic illness.
2. No known renal impairment.
3. 18 Years of age or older at screening.
4. Written informed consent provided by patient or the patient's legally authorized representative.
5. African American and Hispanic participants preferred.

Exclusion Criteria:

1. Recent significant medical condition that required hospitalization (other than sickle cell crisis) within 2 months prior to starting L-glutamine therapy.
2. History of chronic kidney disease Stage 4 (glomerular filtration rate [GFR]=15-29) or Stage 5 (GFR<15 mL/min/1.73 m2).
3. History of chronic liver disease Child Pugh class C (10-15 points).
4. Received any blood products 3 months prior to starting L-glutamine therapy.
5. Currently pregnant or lactating or planning to conceive during the study period.
6. Currently taking or has taken any form of glutamine supplement within 30 days prior to starting L-glutamine therapy.
7. Has been treated with an investigational medication/treatment within 30 days prior to starting L-glutamine therapy.
8. Is currently enrolled in an investigational drug or device study and/or has participated in such a study within 30 days prior to starting L-glutamine therapy.
9. Factors that would, in the judgment of the investigator, make it difficult for the patient to comply with study requirements.
10. Patient is currently being treated with crizanlizumab or voxelotor.

Exclusion Criteria for Healthy Volunteers:

1. Known allergies to L-glutamine.
2. Informed consent document was not completed and signed.
3. Currently pregnant or lactating or planning to conceive during the study period.
4. Known hematologic illness, renal or hepatic impairment.
5. Received any blood products within 3 months of starting L-glutamine therapy.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of L-glutamine at 0.1 g/kg twice daily, 0.3 g/kg twice daily, and 0.6 g/kg once daily in SCD patients | Week 1 Day 1 (0.1 g/kg dose) and Week 2 Day 1 (0.3 g/kg dose. Week 3 Day 1 and Week4 Day1 (0.6 g/kg once daily dose)
  PK (AUC)
Maximum Plasma Concentration (Cmax) of L-glutamine at 0.1 g/kg twice daily, 0.3 g/kg twice daily, and 0.6 g/kg once daily in SCD patients | Week 1 Day 1 (0.1 g/kg dose) and Week 2 Day 1 (0.3 g/kg dose. Week 3 Day 1 and Week4 Day1 (0.6 g/kg once daily dose)
  PK (Cmax)
Half-life (t1/2) of L-glutamine at 0.1 g/kg twice daily, 0.3 g/kg twice daily, and 0.6 g/kg once daily in SCD patients | Week 1 Day 1 (0.1 g/kg dose) and Week 2 Day 1 (0.3 g/kg dose. Week 3 Day 1 and Week4 Day1 (0.6 g/kg once daily dose)
  PK (t1/2)
Time to Peak Concentration (Tmax) of L-glutamine at 0.1 g/kg twice daily, 0.3 g/kg twice daily, and 0.6 g/kg once daily in SCD patients | Week 1 Day 1 (0.1 g/kg dose) and Week 2 Day 1 (0.3 g/kg dose. Week 3 Day 1 and Week4 Day1 (0.6 g/kg once daily dose)
  PK (Tmax)

SECONDARY OUTCOMES:
Glutamate levels | Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, Week 4 Day 1.
  Plasma and serum glutamate levels.
Effect of Food on L-glutamine Area Under Curve (AUC) | Week 1 Day 1, Week 2 Day 1, Week 4 Day 1.
  Food effect on AUC.
Effect of Food on L-glutamine Maximum Plasma Concentration (Cmax) | Week 1 Day 1, Week 2 Day 1, Week 4 Day 1.
  Food effect on Cmax.
L-glutamine Dose Effect on Area Under Curve (AUC) | Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, Week 4 Day 1.
  Dose effect on AUC.
L-glutamine Dose Effect on Maximum Plasma Concentration (Cmax) | Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, Week 4 Day 1.
  Dose effect on Cmax.
L-glutamine Interpatient Variability of Area Under Curve (AUC) | Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, Week 4 Day 1.
  Interpatient variability of AUC.
L-glutamine Interpatient Variability of Maximum Plasma Concentration (Cmax) | Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, Week 4 Day 1.
  Interpatient variability of Cmax.
Ammonia levels | Week 1 Day 1, Week 2 Day 1, Week 3 Day 1, Week 4 Day 1.
  Basal whole blood ammonia levels.

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Niihara, MD, Study Chair — Emmaus Medical, Inc.
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sadaf A, Dong M, Pfeiffer A, Latham T, Kalfa T, Vinks AA, Ware RE, Quinn CT. A Population Pharmacokinetic Analysis of L-Glutamine Exposure in Patients with Sickle Cell Disease: Evaluation of Dose and Food Effects. Clin Pharmacokinet. 2024 Mar;63(3):357-365. doi: 10.1007/s40262-024-01349-4. Epub 2024 Feb 24. PMID 38401036